CLINICAL TRIAL: NCT02811809
Title: Apalutamide Plus Intermittent Hormone Therapy (IHT) Versus IHT Alone in Prostate Cancer Patients With Biochemical Recurrence
Brief Title: Apalutamide Plus Intermittent Hormone Therapy Versus Intermittent Hormone Therapy Alone in Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn due to operational issues. The study was withdrawn early, before enrolling its first participant.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GU-15-105; HSC-MS-16-0477 (Other: CPHS)
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Apalutamide; IHT; BCR; Biochemical recurrence; intermittent hormone therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Apalutamide + IHT (Experimental): Participants will be treated with 240 mg (4-60 mg tablets) oral Apalutamide daily plus 22.5 mg 3-month depot intramuscular leuprolide intermittently.
  Interventions: Drug: Apalutamide; Drug: IHT
- IHT only (Active Comparator): Participants will receive 22.5 mg 3-month depot intramuscular leuprolide until PSA progression, then they will crossover to Apalutamide + IHT
  Interventions: Drug: IHT

INTERVENTIONS:
Drug: Apalutamide — Apalutamide 240 mg (4 60mg tablets) daily
  Other Names: ARN-509; JNJ-56021927
  Arms: Apalutamide + IHT
Drug: IHT — Leuprolide 3-month depot 22.5 intramuscular dose
  Other Names: Leuprolide; Lupron Depot

SUMMARY:
This study is open to men who have biochemical recurrence (BCR, increased PSA) following local treatment of their prostate cancer. Androgen deprivation therapy (ADT) is a standard treatment option, but is only effective for 16-24 months and has a number of side effects that impact quality of life. These side effects may include fatigue, hot flushing, loss of sex drive, brain fog, decreased bone mineral density, loss of muscle mass, mild anemia (low levels of red blood cells that can make people feel tired and weak), diabetes (low blood sugar), heart disease, metabolic syndromes (sometimes called "pre-diabetes" and includes obesity, increased blood pressure, high levels of cholesterol and triglycerides in blood), and risk of fractures. An alternative to continuous ADT is intermittent administration, where patients are given "breaks" from ADT to let their testosterone levels return to baseline. There are a number of potential benefits to intermittent hormone therapy (IHT): (1) longer time to the development of resistance; (2) improved patient quality of life owing to recovery from adverse effects, particularly sexual function; and (3) substantial cost savings owing to less time spent receiving medication. Leuprolide is the name of the ADT / IHT drug.

Apalutamide is an investigational drug, which means it has not been approved by the Food and Drug Administration (FDA). It is an antitumor drug, taken by mouth. The purpose of this study is to determine the ability of Apalutamide to extend the time between the first two injections of leuprolide and improve quality of life. This study will also look at the safety of Apalutamide and the effects that Apalutamide has on prostate cancer.

Men will be randomized (like flipping a coin) to receive:

* Group A: Leuprolide + Apalutamide or
* Group B: Leuprolide only (until second leuprolide injection), then leuprolide + Apalutamide 45 men will be in Group A and 21 men will be in Group B. Leuprolide is given as an intramuscular shot that lasts for 3 months intermittently and Apalutamide is taken by mouth (4 tablets) daily. Each cycle is 4 weeks long.

Intermittent treatment with Apalutamide + leuprolide will continue until continuous leuprolide is needed to maintain undetectable PSA levels (i.e., PSA levels rise above undetectable level unless leuprolide is given without pause, every 3 months).

DETAILED DESCRIPTION:
Prostate-specific antigen (PSA) is a sensitive and specific biomarker of prostate tissue. Monitoring of PSA after local treatment for prostate cancer can assist in identifying patients who have only increased PSA (biochemical recurrence [BCR]) despite no symptoms, signs, or evidence of radiographic metastatic disease. This subpopulation of patients are referred to as having "biochemical failure." Androgen deprivation therapy (ADT) is a standard treatment option, but is only effective for 16-24 months and has a number of side effects that impact quality of life. These side effects may include fatigue, hot flushing, loss of sex drive, brain fog, decreased bone mineral density, loss of muscle mass, mild anemia, diabetes, heart disease, metabolic syndromes and risk of fractures. An alternative to continuous ADT is intermittent administration, where patients are given "breaks" from ADT to let their testosterone levels return to baseline. There are a number of potential benefits to intermittent hormone therapy (IHT): (1) longer time to the development of resistance, owing to the removal of constant pressure causing faster mutation of resistant cells; (2) improved patient quality of life owing to recovery from adverse effects, particularly sexual function; and (3) substantial cost savings owing to less time spent receiving medication. Leuprolide is the name of the ADT / IHT drug.

Apalutamide is an investigational antitumor drug, taken by mouth. It is a synthetic compound rationally designed to bind the androgen receptor (with higher affinity than enzalutamide or bicalutamide), prevent both nuclear translocation and DNA binding, and induce apoptosis. It has greater antitumor activity at a lower dose, achieves steady-state levels at a lower dose, and accumulates more into tumor tissue without building up in the brain, which both increases effectiveness and decreases the risk of seizure.

Apalutamide's mechanism of action gives it the potential to extend the time to PSA increase during intermittent ADT, delaying the necessity for continuous ADT. Investigators will assess the potential applications of intermittent ADT plus Apalutamide for participants with BCR. This study will elucidate the potential of this regimen to reduce the burden of adverse events of continuous ADT and delay the development of hormone resistance.

This is a randomized crossover study intended to determine the interval of ADT administration achievable with supportive Apalutamide treatment. Investigators will assess the significance of time to PSA recurrence, time to next leuprolide injection, time to testosterone recovery, duration of testosterone recovery, time to biochemical recurrence, percentage of men developing biochemical recurrence, number of detectable CTCs, and quality of life measures.

Treatment will be 66 participants in 2:1 randomized crossover - 45 IHT + apalutamide:21 IHT only until second leuprolide injection, then IHT + apalutamide

Apalutamide + IHT Participants will be treated with 240 mg (4 60 mg tablets) oral Apalutamide daily plus 22.5 mg 3-month depot intramuscular leuprolide intermittently.

IHT Participants will receive 22.5 mg 3-month depot intramuscular leuprolide until PSA progression, when they will receive 240 mg oral Apalutamide daily plus 22.5 mg 3-month depot intramuscular leuprolide intermittently.

Participants remain on study until continuous ADT is required to maintain castrate PSA levels (i.e., leuprolide is needed every 3 months to maintain PSA <1 ng/dL).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with a diagnosis of adenocarcinoma of the prostate
* Patients with BCR (PSA becomes detectable, with absolute value ≥1) following prostatectomy who have no evidence of metastatic disease based on radiographic assessment.
* Patients with BCR following radiation therapy who have no radiographic involvement per mpMRI and CT (RTOG-ASTRO Phoenix criteria), size of pelvic nodes ≤1 cm, and whose MRI-directed prostate biopsies are negative.
* Patients must be free of serious comorbidity as determined by investigator.
* Clinical laboratory values at screening:
* Serum testosterone level ≥150 ng/dL
* Hemoglobin ≥9.0 g/dL, independent of transfusion and/or growth factors within 3 months prior to randomization
* Platelet count ≥100,000 /µL independent of transfusion and/or growth factors within 3 months prior to randomization
* Serum albumin ≥3.0 g/dL
* GFR >45 mL/min
* Serum potassium ≥3.5 mmol/L
* Serum total bilirubin ≤1.5 × ULN (Note: In subjects with Gilbert's syndrome, if total bilirubin is >1.5 × ULN, measure direct and indirect bilirubin and if direct bilirubin is ≤1.5 × ULN, subject may be eligible)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) <2.5 × ULN
* Medications known to lower the seizure threshold (see list under prohibited meds, Appendix 3) must be discontinued or substituted at least 4 weeks prior to study entry.
* Agrees to use a condom (even men with vasectomies) and another effective method of birth control if he is having sex with a woman of childbearing potential or agrees to use a condom if he is having sex with a woman who is pregnant while on study drug and for 3 months following the last dose of study drug. Must also agree not to donate sperm during the study and for 3 months after receiving the last dose of study drug.
* Written, informed consent to participate in this study.

Exclusion Criteria:

* PSA doubling time >12 months
* Positive for HIV or chronic hepatitis B or hepatitis C infection
* Another primary malignancy that has not been in remission for at least 2 years. Non-melanoma skin cancer allowed.
* Use of herbal products that may decrease PSA levels (e.g., saw palmetto) or systemic corticosteroids greater than the equivalent of 10 mg of prednisone per day within 4 weeks of screening laboratory studies.
* Any other condition, including concurrent medical condition, social circumstance or drug dependency, which in the opinion of the investigator could compromise patient safety and/or compliance with study requirements
* History of any of the following:

  * Seizure or known condition that may pre-dispose to seizure (e.g. prior stroke within 1year to randomization, brain arteriovenous malformation, Schwannoma, meningioma, or other benign CNS or meningeal disease which may require treatment with surgery or radiation therapy)
  * Severe or unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events (eg, pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or clinically significant ventricular arrhythmias within 6 months prior to randomization Any condition that in the opinion of the investigator, would preclude participation in this study
* Current evidence of any of the following:

  * Uncontrolled hypertension
  * Gastrointestinal disorder affecting absorption
  * Active infection (eg, human immunodeficiency virus [HIV] or viral hepatitis) Any condition that in the opinion of the investigator, would preclude participation in this study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Time to second injection | 48 months
  Time to second injection

SECONDARY OUTCOMES:
Time to prostate-specific antigen (PSA) nadir | 48 months
  Time to prostate-specific antigen (PSA) nadir
Duration of PSA nadir | 48 months
  Duration of PSA nadir
Time to testosterone recovery to >50 ng/dl | 48 months
  Time to testosterone recovery to >50 ng/dl
Duration of testosterone recovery | 48 months
  Duration of testosterone recovery
Circulating tumor cell (CTC) enumeration | 48 months
  Circulating tumor cell (CTC) enumeration
Time until BCR after discontinuation of Apalutamide and ADT | 48 months
  Time until BCR after discontinuation of Apalutamide and ADT
Quality of life as determined by FACT-P survey | 48 months
  Quality of life as determined by FACT-P survey
Number of Adverse Events | 48 months
  Number of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Amato, DO, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- UTHealth Memorial Hermann Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No